CLINICAL TRIAL: NCT00160641
Title: A Phase III Multi-center, Open-label, Follow-up Study, to Assess the Safety and Efficacy of Liquid Certolizumab Pegol as Additional Medication to Methotrexate, in the Treatment of Signs and Symptoms and in the Prevention of Joint Damage in Patients With Active Rheumatoid Arthritis Who Participated in Study CDP870-050
Brief Title: A Study of the Safety and Effectiveness of Liquid Certolizumab Pegol in the Treatment of Signs and Symptoms of Rheumatoid Arthritis and in Prevention of Joint Damage in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87051; 2005-002629-30 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; CDP870; Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab Pegol (Experimental): All patients received Certolizumab Pegol (CZP) 400 mg subcutaneously (sc) every two weeks, given as two 1 ml injections of CZP for at least six months and then 200 mg of CZP sc every two weeks, given as one 1 ml injection.
  Interventions: Biological: Certolizumab Pegol

INTERVENTIONS:
Biological: Certolizumab Pegol — Strength and Form: 1 ml of Liquid product containing 200 mg of Certolizumab Pegol (CZP) given as a subcutaneous injection.
  Dosage and Frequency: 400 mg every two weeks for at least 6 months, then 200 mg every two weeks.
  Duration: Until end of study.
  Other Names: Cimzia

SUMMARY:
An open ended study in which patients who completed the preceding double-blind study NCT00160602 are given Certolizumab Pegol and assessed for signs and symptoms of Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

Patients must have either failed to achieve an American College of Rheumatology 20 % (ACR20) response at Weeks 12 and 14 in C87050 [NCT00160602], or must have completed the entire Week 24 assessment of C87050 [NCT00160602] trial.

Exclusion Criteria:

* A diagnosis of any other inflammatory Arthritis (e.g. Psoriatic Arthritis or Ankylosing Spondylitis)
* A secondary, non-inflammatory type of Arthritis (e.g. Osteoarthritis or Fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of CDP870 on the patient's primary diagnosis of Rheumatoid Arthritis (RA)
* Any concomitant biological therapy
* Any experimental therapy, within or outside a clinical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2005-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (67):
- United States (12):
  - 172, Palm Desert, California
  - 185, Pasadena, California
  - 170, Santa Maria, California
  - 194, Whittier, California
  - 176, Naples, Florida
  - 186, Palm Harbor, Florida
  - 188, Kansas City, Missouri
  - 182, St Louis, Missouri
  - 178, Stratford, New Jersey
  - 192, Amarillo, Texas
  - 173, Austin, Texas
  - 175, San Antonio, Texas
- Bulgaria (2):
  - 303, Pleven
  - 302, Sofia
- 500, Rijeka, Croatia
- Czechia (7):
  - 600, Brno
  - 603, Hlučín
  - 605, Prague
  - 606, Prague
  - 604, Sokolov
  - 602, Uherské Hradiště
  - 607, Zlín
- 700, Tallinn, Estonia
- Israel (6):
  - 802, Afula
  - 805, Ashkelon
  - 807, Haifa
  - 804, Jerusalem
  - 801, Ramat Gan
  - 806, Ẕerifin
- Latvia (2):
  - 901, Daugavpils
  - 900, Riga
- Lithuania (4):
  - 103, Alytus
  - 100, Kaunas
  - 102, Klaipėda
  - 101, Šiauliai
- Poland (6):
  - 124, Bialystok
  - 120, Elblag
  - 123, Krakow
  - 125, Lublin
  - 121, Sopot
  - 122, Torun
- Russia (9):
  - 150, Moscow
  - 151, Moscow
  - 156, Moscow
  - 159, Moscow
  - 152, Saint Petersburg
  - 154, Saint Petersburg
  - 155, Saint Petersburg
  - 158, Saint Petersburg
  - 153, Yaroslavl
- Serbia (3):
  - 132, Belgrade
  - 133, Belgrade
  - 131, Niška Banja
- Slovakia (4):
  - 141, Košice
  - 143, Košice
  - 140, Piešťany
  - 142, Piešťany
- Ukraine (10):
  - 162, Dnipro
  - 161, Donetsk
  - 168, Donetsk
  - 165, Ivano-Frankivsk
  - 163, Kiev
  - 164, Kiev
  - 167, Kiev
  - 169, Kiev
  - 160, Simferopol
  - 166, Zaporizhzhya

REFERENCES:
- [Background] Paul S, Marotte H, Kavanaugh A, Goupille P, Kvien TK, de Longueville M, Mulleman D, Sandborn WJ, Vande Casteele N. Exposure-Response Relationship of Certolizumab Pegol and Achievement of Low Disease Activity and Remission in Patients With Rheumatoid Arthritis. Clin Transl Sci. 2020 Jul;13(4):743-751. doi: 10.1111/cts.12760. Epub 2020 Apr 1. PMID 32100960
- [Derived] Curtis JR, Winthrop K, O'Brien C, Ndlovu MN, de Longueville M, Haraoui B. Use of a baseline risk score to identify the risk of serious infectious events in patients with rheumatoid arthritis during certolizumab pegol treatment. Arthritis Res Ther. 2017 Dec 15;19(1):276. doi: 10.1186/s13075-017-1466-y. PMID 29246162
- [Derived] Smolen JS, van Vollenhoven R, Kavanaugh A, Strand V, Vencovsky J, Schiff M, Landewe R, Haraoui B, Arendt C, Mountian I, Carter D, van der Heijde D. Certolizumab pegol plus methotrexate 5-year results from the rheumatoid arthritis prevention of structural damage (RAPID) 2 randomized controlled trial and long-term extension in rheumatoid arthritis patients. Arthritis Res Ther. 2015 Sep 10;17(1):245. doi: 10.1186/s13075-015-0767-2. PMID 26353833
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started in December 2005. 67 centers in 13 countries enrolled subjects. Participant Flow refers to the Safety Set (SS) consisting of all enrolled subjects who received at least 1 dose of study medication. Due to fraud findings at 1 site, data of the 15 subjects of site were not analyzed with data from all other sites and not part of SS.
Pre-assignment Details: This Open-label Study consists of two different populations:
  of those subjects who failed to achieve predefined criteria in preceding study C87050 [NCT00160602] who entered C87051 on Week 16 of the preceding study and of those who completed the Week 24 assessment of the preceding study.
Groups:
- Certolizumab Pegol: All patients received Certolizumab Pegol (CZP) 400 mg subcutaneously (sc) every two weeks, given as two 1 ml injections of CZP for at least six months and then 200 mg of CZP sc every two weeks, given as one 1 ml injection.
  Certolizumab Pegol : Strength and Form: 1 ml of Liquid product containing 200 mg of Certolizumab Pegol (CZP) given as a subcutaneous injection.
  Dosage and Frequency: 400 mg every two weeks for at least 6 months, then 200 mg every two weeks.
  Duration: Until end of study.
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 567
Completed | 346
Not Completed | 221
Not completed — Adverse Event | 102
Not completed — Withdrawal by Subject | 87
Not completed — Lost to Follow-up | 8
Not completed — Lack of Efficacy | 12
Not completed — Protocol Violation | 3
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS). SS consists of all enrolled subjects who received at least 1 dose of study medication.
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 567
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 486
  >=65 years | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 463
  Male | 104
Region of Enrollment [Number; unit: participants]
  United States | 35
  Serbia | 46
  Estonia | 6
  Slovakia | 30
  Ukraine | 70
  Lithuania | 43
  Israel | 17
  Russian Federation | 105
  Czech Republic | 93
  Poland | 86
  Croatia | 10
  Bulgaria | 14
  Latvia | 12
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 72.37 (14.86)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 165.23 (8.16)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Adverse Event (AE) From First Certolizumab Pegol (CZP) Dose up to Approximately 6.8 Years
Description: An AE is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage. First dose of CZP was at Baseline of the preceding double-blind study NCT00160602 for subjects randomized to CZP, or at Entry Visit (Week 0) of this study for subjects randomized to Placebo.
Time Frame: From first dose of CZP to the end of the open-label study (approximately 6.8 years)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 567
percentage of participants | 89.1

2. Primary Outcome: Percentage of Subjects With at Least One Serious Adverse Event (SAE) From First Certolizumab Pegol (CZP) Dose up to Approximately 6.8 Years
Description: A SAE is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly or birth defect
  * Is as infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above
  First dose of CZP was at Baseline of the preceding double-blind study NCT00160602 for subjects randomized to CZP, or at Entry Visit (Week 0) of this study for subjects randomized to Placebo.
Time Frame: From first dose of CZP to the end of the open-label study (approximately 6.8 years)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 567
percentage of participants | 35.3

3. Primary Outcome: Percentage of Subjects Who Withdrew Due to an Adverse Event (AE) During the Study
Description: An AE is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device.
  The event does not necessarily have a causal relationship with that treatment or usage. The results of this Primary Outcome Measure are summarized from the Adverse Event pages of the Case Report Forms.
Time Frame: From Entry Visit (Week 0) to the end of the study (approximately 6.3 years)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 567
percentage of participants | 17.6

4. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 52
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 52 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 52 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 493 are included in this analysis. Data not available for 74 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 493
percentage of participants | 81.7 [78.0 to 85.1]

5. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 100
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 100 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 100 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 442 are included in this analysis. Data not available for 125 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 442
percentage of participants | 79.4 [75.3 to 83.1]

6. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 148
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 148 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 148 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 410 are included in this analysis. Data not available for 157 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 410
percentage of participants | 80.2 [76.1 to 84.0]

7. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 196
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 196 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 196 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 367 are included in this analysis. Data not available for 200 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 367
percentage of participants | 81.5 [77.1 to 85.3]

8. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 244
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 244 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 244 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 72 are included in this analysis. Data not available for 495 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 72
percentage of participants | 88.9 [79.3 to 95.1]

9. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Completion/Withdrawal
Description: The assessments are based on a 20 % or greater improvement from Baseline to Completion/Withdrawal in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Completion/Withdrawal of the open-label study (up to approximately 6.8 years)
Population: Of the 567 subjects in the Safety Set (SS), 565 are included in this analysis. Data not available for 2 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 565
percentage of participants | 74.2 [70.3 to 77.7]

10. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 52
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 52 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 52 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 493 are included in this analysis. Data not available for 74 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 493
percentage of participants | 48.9 [44.4 to 53.4]

11. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 100
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 100 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 100 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 442 are included in this analysis. Data not available for 125 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 442
percentage of participants | 51.4 [46.6 to 56.1]

12. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 148
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 148 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 148 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 410 are included in this analysis. Data not available for 157 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 410
percentage of participants | 51.7 [46.8 to 56.6]

13. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 196
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 196 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 196 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 367 are included in this analysis. Data not available for 200 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 367
percentage of participants | 56.9 [51.7 to 62.1]

14. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 244
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 244 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 244 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 72 are included in this analysis. Data not available for 495 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 72
percentage of participants | 62.5 [50.3 to 73.6]

15. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Completion/Withdrawal
Description: The assessments are based on a 50 % or greater improvement from Baseline to Completion/Withdrawal in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: as for outcome 9
Population: Of the 567 subjects in the Safety Set (SS), 565 are included in this analysis. Data not available for 2 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 565
percentage of participants | 47.4 [43.3 to 51.6]

16. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 52
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 52 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 52 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 493 are included in this analysis. Data not available for 74 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 493
percentage of participants | 26.2 [22.3 to 30.3]

17. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 100
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 100 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 100 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 442 are included in this analysis. Data not available for 125 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 442
percentage of participants | 27.1 [23.1 to 31.6]

18. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 148
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 148 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 148 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 410 are included in this analysis. Data not available for 157 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 410
percentage of participants | 25.6 [21.5 to 30.1]

19. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 196
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 196 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 196 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 367 are included in this analysis. Data not available for 200 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 367
percentage of participants | 29.4 [24.8 to 34.4]

20. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 244
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 244 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 244 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 72 are included in this analysis. Data not available for 495 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 72
percentage of participants | 31.9 [21.4 to 44.0]

21. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Completion/Withdrawal
Description: The assessments are based on a 70 % or greater improvement from Baseline to Completion/Withdrawal in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: as for outcome 9
Population: Of the 567 subjects in the Safety Set (SS), 565 are included in this analysis. Data not available for 2 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 565
percentage of participants | 25.5 [21.9 to 29.3]

22. Secondary Outcome: Change From Baseline of the Preceding Double-Blind Study to Week 104 in Modified Total Sharp Score (mTSS)
Description: The mTSS quantifies the extent of bone erosions and joint space narrowing for 44 and 42 joints, respectively, as assessed by x-rays of the hands and feet. The score ranges from 0 to 448 with higher scores representing greater damage. A negative value in mTSS change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: From Baseline of the preceding double-blind study to Week 104 of the open-label study
Population: Of the 567 subjects in the Safety Set (SS), 423 are included in this analysis. Data not available for 144 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 423
units on a scale | 0.99 (4.99)

23. Secondary Outcome: Change From Baseline of the Preceding Double-Blind Study to Completion/Withdrawal Visit in Health Assessment Questionnaire - Disability Index (HAQ-DI) Total Score
Description: The HAQ-DI assesses the degree of difficulty experienced in eight domains (Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Gripping, Other Activities) of daily living activities using 20 questions. The HAQ-DI is calculated by summing the domain scores and dividing them by the number of domains. It ranges from 0 (no difficulty) to 3 (unable to do). Negative values indicate an improvement from Baseline to the Post-Baseline Visit with larger negative values showing a better improvement.
Time Frame: as for outcome 9
Population: Of the 567 subjects in the Safety Set (SS), 560 are included in this analysis. Data not available for 7 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 560
units on a scale | -0.567 (0.633)

24. Secondary Outcome: Change From Baseline to Completion/Withdrawal Visit in Duration of Morning Stiffness
Description: Morning stiffness is defined as the time in hours elapsed between the time of usual awakening (even if not in the morning) and the time the subject is as limber as he/she will be during a day involving typical activities. A negative value in duration of morning stiffness change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: as for outcome 9
Population: Of the 567 subjects in the Safety Set (SS), 563 are included in this analysis. Data not available for 4 subjects.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 563
hours | -2.31 (3.31)

25. Secondary Outcome: Change From Baseline to Completion/Withdrawal Visit in Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28[ESR])
Description: DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/ hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. A negative value in DAS28[ESR] change from Baseline indicates an improvement from Baseline.
Time Frame: as for outcome 9
Population: Of the 567 subjects in the Safety Set (SS), 556 are included in this analysis. Data not available for 11 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 556
units on a scale | -2.990 (1.408)

26. Secondary Outcome: Percentage of Subjects With Good European League Against Rheumatism (EULAR) Response at Completion/Withdrawal Visit
Description: Good EULAR response is defined as DAS28[ESR] improvement from Baseline of the preceding double-blind study > 1.2 and DAS28[ESR] value < 3.2.
Time Frame: as for outcome 9
Population: Of the 567 subjects in the Safety Set (SS), 556 are included in this analysis. Data not available for 11 subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 556
percentage of participants | 36.0

27. Secondary Outcome: Change From Baseline to Completion/Withdrawal Visit in Short-Form Health Survey (SF-36) Item Questionnaire Physical Component Summary (PCS) Score
Description: The SF-36 is a 36-item generic health status measure that measures 8 general health concepts: Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each domain of the eight domains and the summary concept PCS score are scored to yield values between 0 (worst) and 100 (best).
Time Frame: as for outcome 9
Population: Of the 567 subjects in the Safety Set (SS), 527 are included in this analysis. Data not available for 40 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 527
units on a scale | 6.628 (8.950)

28. Secondary Outcome: Change From Baseline to Completion/Withdrawal Visit in Short-Form Health Survey (SF-36) Item Questionnaire Mental Component Summary (MCS) Score
Description: The SF-36 is a 36-item generic health status measure that measures 8 general health concepts: Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each domain of the eight domains and the summary concept MCS score are scored to yield values between 0 (worst) and 100 (best).
Time Frame: as for outcome 9
Population: Of the 567 subjects in the Safety Set (SS), 527 are included in this analysis. Data not available for 40 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 527
units on a scale | 4.325 (12.208)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to approximately 6.8 years, from first dose of Certolizumab Pegol (CZP) to the end of the open-label study.
Description: AEs refer to the Safety Set. Safety Set includes all enrolled subjects who received at least 1 dose of study medication.
Arm/Group | Certolizumab Pegol
Serious Adverse Events (participants affected / at risk) | 200/567
Other Adverse Events (participants affected / at risk) | 383/567
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=567)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4)
Myocardial ischaemia (Cardiac disorders) | 2 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Cataract (Eye disorders) | 2 (2)
Uveitis (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Periproctitis (Gastrointestinal disorders) | 1 (1)
Death and sudden death (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 5 (5)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 5 (5)
Gangrene (Infections and infestations) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Bursitis infective (Infections and infestations) | 3 (3)
Osteomyelitis (Infections and infestations) | 1 (1)
Borrelia infection (Infections and infestations) | 2 (2)
Lyme disease (Infections and infestations) | 1 (1)
Colitis pseudomembranous (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 2 (3)
Salpingo-oophoritis (Infections and infestations) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1)
Gallbladder empyema (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Bronchitis acute (Infections and infestations) | 2 (2)
Bronchopneumonia (Infections and infestations) | 2 (3)
Embolic pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9)
Pneumonia primary atypical (Infections and infestations) | 1 (1)
Papilloma viral infection (Infections and infestations) | 1 (2)
Carbuncle (Infections and infestations) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 3 (3)
Pneumococcal sepsis (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Toxic shock syndrome streptococcal (Infections and infestations) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 1 (1)
Meningitis tuberculous (Infections and infestations) | 1 (2)
Pulmonary tuberculosis (Infections and infestations) | 9 (9)
Tuberculosis (Infections and infestations) | 4 (4)
Tuberculosis of central nervous system (Infections and infestations) | 1 (1)
Tuberculosis of intrathoracic lymph nodes (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Pyelocystitis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 4 (4)
Pyelonephritis chronic (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hernia (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 (7)
Flat feet (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower limb deformity (Musculoskeletal and connective tissue disorders) | 1 (2)
Toe deformity (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (11)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 19 (22)
Fistula (Musculoskeletal and connective tissue disorders) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Acoustic neuritis (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Radicular syndrome (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 7 (9)
Vocal cord paralysis (Nervous system disorders) | 1 (2)
Mental disorder (Psychiatric disorders) | 1 (1)
Glomerulonephritis proliferative (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 3 (4)
Ovarian cyst (Reproductive system and breast disorders) | 4 (4)
Colpocele (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 (2)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Peritoneal adhesions division (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 2 (2)
Varicose ulceration (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=567)
Upper respiratory tract infection (Infections and infestations) | 91 (150)
Nasopharyngitis (Infections and infestations) | 65 (99)
Urinary tract infection (Infections and infestations) | 60 (90)
Bronchitis acute (Infections and infestations) | 52 (69)
Viral infection (Infections and infestations) | 46 (61)
Pharyngitis (Infections and infestations) | 33 (48)
Respiratory tract infection (Infections and infestations) | 31 (48)
Activated partial thromboplastin time prolonged (Investigations) | 65 (106)
Alanine aminotransferase increased (Investigations) | 29 (42)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 76 (146)
Back pain (Musculoskeletal and connective tissue disorders) | 44 (56)
Headache (Nervous system disorders) | 44 (61)
Hypertension (Vascular disorders) | 77 (85)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days